CLINICAL TRIAL: NCT06709235
Title: Characterization of Infectious Events and Their Impact on Survival in Patients with Acute Myeloid Leukemia Treated with Intensive Chemotherapy
Brief Title: Assessing Refractoriness and Infectious Survival Events in AML
Acronym: ARISE-AML
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 23-5053
Record Dates: First submitted 2024-11-21; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Acute myeloid leukemia; infections; intensive chemotherapy; survival
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- AML patients treated with intensive chemotherapy: Patients diagnosed with acute myeloid leukemia treated in our center with 3+7 based induction chemotherapy regimen

SUMMARY:
Despite therapeutic advance in acute myeloid leukemia (AML), the prognosis remains poor, with an overall survival (OS) of 30% at 5 years [1, 2]. Treatment of 1st-line AML in patients under 75 years of age is based on intensive chemotherapy (IC) followed by allogeneic transplantation (hematopoietic stem cell transplantation, HSCT) [3]. Following its administration, a phase known as aplasia ensues, during which patients are severely immunocompromised. This period of aplasia therefore carries a very high risk of infectious events, despite management in protected areas and infectious prophylaxis. Infectious problems remain one of the leading causes of mortality in the initial phase of AML treatment [4]. The incidence of sepsis, the microorganisms involved and the complications arising from infectious episodes during chemotherapy remain poorly described, as do their long-term prognostic consequences for these patients [5,6].

Moreover, there is a "dogma" among hematologists dealing specifically with AML that intensive chemotherapy during which there are no infectious events is often a sign of non-response. Although this "popular" belief has never been verified prospectively or even retrospectively, it is based on the observation of many generations of clinicians. This belief suggests that immune stimulation during aplasie could promote remission by inducing an anti-leukemic immune response. Furthermore, numerous cases of "spontaneous" remission (i.e. in AML patients receiving no active treatment) following infections or highly immune-stimulating events have been reported in the literature [7-10].

It might therefore be hypothesized that infectious events occurring during the post-intensive chemotherapy aplasia phase for AML could favor the achievement of remission by nonspecific immune stimulation.

The aim of this study is to describe the incidence and type of septic episodes occurring in patients undergoing intensive treatment for acute myeloid leukemia, and to assess the impact of these episodes on patient prognosis, notably via the risk of relapse and long-term survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute myeloid leukemia (AML)
* Age over 18 years
* Treatment with "intensive" chemotherapy (combination of aracytin and an anthracycline)
* Date of diagnosis of acute myeloid leukemia between 01/01/2015 and 31/12/2021
* Treatment received at Hospices Civils de Lyon (HCL)

Exclusion Criteria:

* Patients with acute promyelocytic leukemia (AML 3)
* Treatment with "non-intensive" chemotherapy (i.e. azacytidine)
* Death before first post-chemotherapy bone marrow assessment
* No computerized data available
* Follow-up at a center other than HCL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an AML diagnosis during the screening period (01/01/2015 and 31/12/2021) receiving intensive chemotherapy and evaluable at the end of induction phase.
Sampling Method: Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Description of the incidence, nature and complications engendered by the occurrence of infectious events during intensive management for AML. | through study completion, during 3 mounths
  Analysis of the number, type, and complications of infectious events observed during the induction and consolidation phases of intensive management for AML.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Lyon Sud, Pierre-Bénite, France